CLINICAL TRIAL: NCT06938386
Title: Haskap Berry Derived Plasma Metabolites - Pilot Timing Project
Brief Title: Pilot Haskap Metabolite Timing Project
Acronym: PHMTiming
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montana State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2024-2029
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Microbial Colonization; Metabolic Disease; Digestion
Keywords: Polyphenols; Plasma metabolome; Microbial Metabolism; Metabolomics
MeSH Terms: conditions — Communicable Diseases; Metabolic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Haskap (Experimental): Haskap puree will be consumed by all participants after a fasting blood sample is collected
  Interventions: Dietary Supplement: Haskap

INTERVENTIONS:
Dietary Supplement: Haskap — A whole, frozen Haskap berry puree blended with water in a 2:1 ratio of berry to water.

SUMMARY:
Diet is a key factor in managing health and individuals at risk of developing metabolic syndrome or other chronic diseases have the opportunity to use diet as a tool to improve their health. This can be complicated when considering the numerous variables that impact digestion and absorption of key health-promoting compounds in foods. One of these variables is the gut microbiome, a microbial community in the digestive tract that interacts with the foods we consume. The mechanisms the microbiome uses to interact with bioactive compounds in foods, like polyphenols, can modulate the health-promoting benefits of polyphenols. Polyphenols are secondary plant metabolites, commonly found in fruit, legumes, chocolate, coffee, and nuts among other foods that have been shown to improve cardiovascular and metabolic health, as well as reduce inflammation and oxidative stress.

DETAILED DESCRIPTION:
Haskap berries (Lonicera caerulea L.), also known as Blue Honeysuckle or Honeyberry, are a polyphenol rich berry that has a greater polyphenolic content than other commonly consumed berries, like strawberries or blueberries. Haskap berries are unique, having a greater content of polyphenols compared to other foods, specifically cyanidin-3-glucoside. Cyanidin-3-glucoside is an anthocyanin shown to reduce inflammation and cardioprotective effects. There is a growing body of literature describing the impact of berry consumption on metabolic health; however, Haskap berry specific investigations in human participants are limited. Currently, Haskap berry consumption shows promising findings in research related to glycemic control, oxidative stress, and inflammation in in-vitro and mice models. The benefits of Haskap berries as a functional food are highly encouraging in animal models, but translational research to demonstrate beneficial health impacts in humans is needed.

A crucial aspect of polyphenol metabolism is the role of the gut microbiome, which influences both metabolic responses to polyphenol consumption and the bioavailability of polyphenolic metabolites. Polyphenol digestion differs based on the structure of the polyphenol and what area of digestive tract is being considered. In the mouth, mastication and salivary enzymes begin the digestion process. However, polyphenols bind with salivary proteins, like tannin-binding salivary proteins, that inhibit their breakdown and subsequent absorption. In the stomach, a limited amount of polyphenols are broken down and/or absorbed and other are conjugated with glucuronic acid. In the small intestine, polyphenols are hydrolyzed into smaller subunits to be absorbed by both passive and active transport. Lastly, the large intestine is the most important segment of digestion to consider.

One of the challenges of polyphenolic research is the intricate relationship between the gut microbiota and the absorption of polyphenolic compounds. Bacteria in the gut are responsible for the majority of polyphenol digestion. Bacteria in the gut interact with polyphenols in a variety of biotransformation reactions including esterification, dehydroxylation, reduction, and decarboxylation. Certain bacteria in the gut have the ability to perform these reactions with polyphenols, including but not limited to Flavonifractor plautii and Bifidobacterium spp. Polyphenol consumption has been shown to modulate microbial composition; however, this project aims to understand how the microbiome impacts metabolite abundance.

This project aims to bridge an important gap that is how the gut microbiome impacts dietary polyphenol absorption and metabolism and how this impacts the health-promoting compounds in Haskap berries. The purpose of this research proposal is to investigate how the microbiome impacts metabolism of polyphenols from Haskap berries. Overarching hypothesis: The composition of bacteria in the gut of participants will impact the Haskap-related metabolites produced

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old
* Body mass index (BMI) between 18-30 kg/m^2

Exclusion Criteria:

* allergy to Haskap berries
* have taken antibiotics in the last 90 days
* take dietary supplements
* have adverse events from blood draws
* take medication to lower cholesterol, inflammation, lipids
* smoke cigarettes
* pregnant and/or lactating
* have diabetes
* are unwilling to follow a no-polyphenolic diet for 10 days

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Metabolite Abundance | 48 hours
  Relative abundance of metabolites and degradation products of Haskap berries
Metabolite Identity | 48 hours
  Identify metabolites with fragmentation MS/MS data

CONTACTS AND LOCATIONS:
Overall Officials: Mary P Miles, PhD, Principal Investigator — Montana State University
Locations (1):
- Montana State University, Bozeman, Montana, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-04-10): https://cdn.clinicaltrials.gov/large-docs/86/NCT06938386/ICF_000.pdf